CLINICAL TRIAL: NCT05084586
Title: Comparison of the Efficacy and Safety of Continuous and Single-Dose Intravesical Epirubicin Instillation in the Early Postoperative Period of Bladder Cancer
Brief Title: Comparison of the Efficacy and Safety of Continuous and Single-Dose Intravesical Epirubicin Instillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BC2021EPI
Record Dates: First submitted 2021-09-02; First posted 2021-10-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer; Epirubicin Adverse Reaction; Superficial Bladder Cancer; Tumor Recurrence
Keywords: Non-Muscle Invasive Bladder Cancer; Epirubicin; Intravesical Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous Intravesical Infusion of Epirubicin (Active Comparator): Patients who received continuous epirubicin infusion into the bladder in the early postoperative period.
  Interventions: Drug: Intravesical Solution
- Single-Dose Instillation of Epirubicin (Sham Comparator): Patients who received single-dose epirubicin into the bladder in the early postoperative period.
  Interventions: Drug: Intravesical Solution

INTERVENTIONS:
Drug: Intravesical Solution — After the Transurethral Resection of Bladder Tumor(TURBT) surgery, 50 mg Epirubicin solution in 150 ml saline was continuously instiled into the bladder for 2 hours. A drainage catheter was closed in order to fill the bladder with epirubicin solution.
  Other Names: Continuous Epirubicin Instillation During the Early Postoperative Period
  Arms: Continuous Intravesical Infusion of Epirubicin
Drug: Intravesical Solution — After the Transurethral Resection of Bladder Tumor(TURBT) surgery, 50 mg Epirubicin solution in 50 ml saline was instiled into the bladder for 2 hours. A drainage catheter was closed in order to fill the bladder with epirubicin solution.
  Other Names: Single-Dose Epirubicin Instillation During the Early Postoperative Period
  Arms: Single-Dose Instillation of Epirubicin

SUMMARY:
In this study, the local and systemic side effects, tumor recurrens and progression rates of single or continuous epirubicin instillation during the early postoperative period were investigated in low and intermediate risk non-muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Bladder cancer (BC) is the seventh most commonly diagnosed cancer in the male population worldwide, while it drops to tenth when both genders are considered. Worldwide, the BC age-standardised mortality rate (per 100,000 person/years) was 3.3 for men vs. 0.86 for women.It is more common, especially in developed countries. NMIBC are divided into four groups as low-medium-high and very high risk according to EORTC (European Organization for Research and Treatment of Cancer).

Epirubicin is an anthracycline drug used for chemotherapy. Immediate single instillation of epirubicin has been shown to act by destroying circulating tumour cells after TURB(Transurethral Resection of a Bladder Tumor), and by an ablative effect on residual tumour cells at the resection site and on small overlooked tumours.European Association of Urology Guidelines on Bladder Cancer advocates single immediate postoperative intravesical chemotherapy. Early single-dose instillation of epirubicin immediately after transurethral resection was shown to improve recurrence rates in low and intermediate risk groups.

Immediate single instillation of epirubicin into the bladder can induce an array of irritative voiding symptoms including dysuria, frequency, urgency, suprapubic discomfort, hematuria and pelvic pain. In some cases, patients cannot tolerate these symptoms and may necessitate removal of chemotherapeutic agent for alleviation. Incomplete instillation leads to an increase in recurrence and progression rates. In this study, continuous infusion of epirubicin into the bladder and instillation of a single dose epirubicin will be evaluated in terms of side effects, tumor recurrence and progression rates.

ELIGIBILITY:
Inclusion Criteria:

* Low and intermediate risk NMIBC

Exclusion Criteria:

* High risk NMIBC
* Patients who received intravesical BCG
* Postoperative gross hematuria
* Bladder perforation
* Pregnancy
* Urinary tract infection
* Epirubicin allergy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-11-05 (Estimated)

PRIMARY OUTCOMES:
Rate of Tumor Recurrence and Progression | 1 year
  Rate of tumor recurrence and progression after intravesical epirubicin therapyepirubicin treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

REFERENCES:
- [Background] Engeler DS, Wyler S, Neyer M, Hobi C, Muller J, Schmid HP. Feasibility of early intravesical instillation chemotherapy after transurethral resection of the bladder: a prospective evaluation in a consecutive series of 210 cases. Scand J Urol Nephrol. 2008;42(6):522-7. doi: 10.1080/00365590802133099. PMID 18609290
- [Background] Maekawa S, Suzuki H, Ohkubo K, Aoki Y, Okada T, Maeda H, Ogura K, Arai Y. [Continuous intravesical instillation of epirubicin immediately after transurethral resection of superficial bladder cancer: a prospective controlled study]. Hinyokika Kiyo. 2000 May;46(5):301-6. Japanese. PMID 10876750
- [Background] Wu ZB, Lin GB, Chen BJ, Wu ZM, Rong RM. [Efficacy and safety of different dosages of intravesical epirubicin instillation for prevention of primary superficial bladder carcinoma from recurrence]. Zhonghua Zhong Liu Za Zhi. 2005 Aug;27(8):507-9. Chinese. PMID 16188156